CLINICAL TRIAL: NCT01195272
Title: A 52 Week, Single Center, Open-label Study to Evaluate Neutrophil Function and Survival Effects of Tocilizumab (TCZ) in Patients With Active Rheumatoid Arthritis (RA) on Background Non-biologic DMARDs Who Have an Inadequate Response to Current Non-biologic DMARD and/or Anti-TNF Therapy
Brief Title: A Study of the Effects of RoActemra/Actemra (Tocilizumab) on Neutrophils in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Biologic and/or Non-biologic DMARDs.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25243; 2010-018331-18
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv every 4 weeks, 52 weeks

SUMMARY:
This open-label, single arm study will assess the effect of RoActemra/Actemra (tocilizumab) on neutrophils and monitor safety and benefit-risk of RoActemra/Actemra treatment in patients with active rheumatoid arthritis who have an inadequate response to current biologic or non-biologic disease-modifying antirheumatic drugs (DMARDs). Patients will receive RoActemra/Actemra at a dose of 8 mg/kg intravenously every 4 weeks, either as monotherapy or in combination with their current non-biologic DMARD. Anticipated time on study treatment is 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Moderate to severe active rheumatoid arthritis of >/= 6 months duration
* DAS28 >/= 3.2 at screening and baseline
* Inadequate response to biologic or non-biologic DMARDs
* Biologic DMARDs must be withdrawn (approximately 5 half-lives for the agent) before first dose of study drug
* If continuing on a non-biologic DMARD, dose should be stable for at least 8 weeks
* Oral corticosteroids must have been at stable dose for at least 25 out of 28 days prior to baseline

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to screening or not recovered from prior surgery
* Rheumatic autoimmune disease other then RA
* Functional class IV as defined by the American College of Rheumatology (ACR) classification
* Prior history of or current inflammatory joint disease other than RA
* Previous treatment with any cell-depleting therapies
* Intraarticular or parenteral corticosteroids within 4 weeks prior to baseline
* Active infection or history of recurrent infection
* Positive for HIV or hepatitis B or C
* History of or current primary or secondary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Liverpool, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 Milligrams Per Kilogram (mg/kg): Participants received tocilizumab 8 mg/kg (maximum dose 800 mg) intravenously (IV), once every 4 weeks up to 52 weeks (total of 13 infusions).
Period: Overall Study
Arm/Group | Tocilizumab 8 Milligrams Per Kilogram (mg/kg)
Started | 21
Completed | 17
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of tocilizumab treatment and had at least 1 post-baseline safety assessment.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg (maximum dose 800 mg) IV, once every 4 weeks up to 52 weeks (total of 13 infusions).
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage of Cells Staining Positive for Annexin V Binding in Apoptosis
Description: Aging neutrophils translocate phosphatidylserine from the inner leaflet of the plasma membrane to the outer leaflet during the early stages of apoptosis. This translocation can be measured due to the affinity of fluorescein isothiocyanate (FITC)-labeled annexin V to bind exposed phosphatidylserine. Cells that stain positive to Annexin V binding are apoptotic. At 4 hours (hrs) and 20 hrs stimulated and control samples were analyzed for levels of apoptosis.
Time Frame: Visits 2, 3, 5, and 8 (Baseline and Weeks 4, 12 and 24)
Population: Intent-to-treat (ITT) Population: all participants in the Safety Population who provided follow-up data for neutrophils or at least 1 efficacy variable. n (number) equals (=) number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percentage of cells staining positive
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
percentage of cells staining positive
  Visit 2, 4 hrs (n=19) | 8.95 (5.46)
  Visit 3, 4 hrs (n=19) | 7.36 (4.18)
  Visit 5, 4 hrs (n=19) | 8.45 (4.64)
  Visit 8, 4 hrs (n=15) | 12.43 (6.34)
  Visit 2, 20 hrs (n=19) | 53.97 (8.97)
  Visit 3, 20 hrs (n=19) | 50.32 (10.64)
  Visit 5, 20 hrs (n=19) | 50.50 (15.51)
  Visit 8, 20 hrs (n=15) | 48.24 (10.37)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.308, t-test, 2 sided
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.415, t-test, 2 sided
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.335, t-test, 2 sided
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.120, t-test, 2 sided
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.061, t-test, 2 sided
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.031, t-test, 2 sided
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.131, t-test, 2 sided
Statistical Analysis 8: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.202, t-test, 2 sided
Statistical Analysis 9: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.484, t-test, 2 sided
Statistical Analysis 10: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.047, t-test, 2 sided
Statistical Analysis 11: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.285, t-test, 2 sided
Statistical Analysis 12: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.315, t-test, 2 sided

2. Primary Outcome: Mean Percentage of Cells Staining Positive for Annexin V Binding With Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF)
Description: Aging neutrophils translocate phosphatidylserine from the inner leaflet of the plasma membrane to the outer leaflet during the early stages of apoptosis. This translocation can be measured due to the affinity of FITC-labeled annexin V to bind exposed phosphatidylserine. Cells that stain positive to Annexin V binding are apoptotic. At 4 hrs and 20 hrs stimulated and control samples were analyzed for levels of apoptosis. GM-CSF is an agent that delays apoptosis. Percentage of cells that stained positive for Annexin V binding in the presence or absence of GM-CSF (GM-CSF delayed or constitutive) were determined by flow cytometry.
Time Frame: Visits 2, 3, 5, and 8 (Baseline and Weeks 4, 12 and 24)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percentage of cells staining positive
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
percentage of cells staining positive
  Visit 2, 4 hrs (n=19) | 5.46 (6.73)
  Visit 3, 4 hrs (n=19) | 4.18 (7.13)
  Visit 5, 4 hrs (n=19) | 4.64 (3.18)
  Visit 8, 4 hrs (n=15) | 6.34 (2.58)
  Visit 2, 20 hrs (n=19) | 27.00 (11.16)
  Visit 3, 20 hrs (n=19) | 28.35 (10.95)
  Visit 5, 20 hrs (n=19) | 29.68 (14.78)
  Visit 8, 20 hrs (n=15) | 27.79 (12.01)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.288, t-test, 2 sided
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.318, t-test, 2 sided
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.400, t-test, 2 sided
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.317, t-test, 2 sided
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.137, t-test, 2 sided
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; 4 hrs: Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.052, t-test, 2 sided
Statistical Analysis 7: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.354, t-test, 2 sided
Statistical Analysis 8: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.266, t-test, 2 sided
Statistical Analysis 9: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.378, t-test, 2 sided
Statistical Analysis 10: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.422, t-test, 2 sided
Statistical Analysis 11: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.444, t-test, 2 sided
Statistical Analysis 12: Comparison: Tocilizumab 8 mg/kg; 20 hrs: Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.345, t-test, 2 sided

3. Primary Outcome: Mean Fluorescence Intensity of CD11b on Neutrophil Surface
Description: Neutrophils were incubated with labeled antibodies against CD11b. Flow cytometry was used to determine the mean fluorescence intensity. Greater fluorescence correlates with greater adhesion, migration, and ingestion of complement-opsonized particles.
Time Frame: Visits 2, 3, and 5 (Baseline and Weeks 4 and 12)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: fluorescence intensity unit
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
fluorescence intensity unit
  Visit 2 (n=19) | 286.40 (105.86)
  Visit 3 (n=17) | 275.33 (127.37)
  Visit 5 (n=16) | 240.93 (77.50)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.39, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.08, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.18, ANOVA

4. Primary Outcome: Mean Fluorescence Intensity of CD18 on Neutrophil Surface
Description: Neutrophils were incubated with labeled antibodies against CD18. Flow cytometry was used to determine the mean fluorescence intensity. Greater fluorescence correlates with greater adhesion, migration, and ingestion of complement-opsonized particles.
Time Frame: Visits 2, 3, and 5 (Baseline and Weeks 4 and 12)
Population: ITT Population; n=number of participants analyzed at each visit
Measure: Mean (Standard Deviation); unit: fluorescence intensity unit
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
fluorescence intensity unit
  Visit 2 (n=19) | 20.33 (8.30)
  Visit 3 (n=17) | 20.47 (12.31)
  Visit 5 (n=16) | 22.47 (15.42)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.48, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.30, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.34, ANOVA

5. Primary Outcome: Mean Fluorescence Intensity of CD62L (L Selectin) on Neutrophil Surface
Description: Neutrophils were incubated with labeled antibody against CD62L (L selectin). Flow cytometry was used to determine the mean fluorescence intensity. Greater fluorescence correlates with greater adhesion of neutrophils to vessel walls.
Time Frame: Visits 2, 3 and 5 (Baseline and Weeks 4 and 12)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: fluorescence intensity unit
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
fluorescence intensity unit
  Visit 2 (n=19) | 20.56 (10.05)
  Visit 3 (n=17) | 23.40 (11.55)
  Visit 5 (n=16) | 19.93 (15.32)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.44, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.23, ANOVA

6. Primary Outcome: Mean Fluorescence Intensity of CD63 on Neutrophil Surface
Description: Neutrophils were incubated with labeled antibody against CD63b. Flow cytometry was used to determine the mean fluorescence intensity. Greater fluorescence correlates with greater azurophilic degranulation, an indicator of greater microbe killing.
Time Frame: Visits 2, 3, and 5 (Baseline and Weeks 4 and 12)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: fluorescence intensity unit
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
fluorescence intensity unit
  Visit 2 (n=19) | 31.00 (20.68)
  Visit 3 (n=17) | 26.34 (14.55)
  Visit 5 (n=16) | 30.28 (16.53)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.46, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.24, ANOVA

7. Primary Outcome: Mean Fluorescence Intensity of Interleukin-6 Receptor (Il-6R) on Neutrophil Surface
Description: Neutrophils were incubated with labeled antibody against IL-6R. Flow cytometry was used to determine the mean fluorescence intensity. Greater fluorescence correlates with greater density of membrane bound IL-6 receptor.
Time Frame: Visits 2, 3, and 5 (Baseline and Weeks 4 and 12)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: fluorescence intensity unit
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
fluorescence intensity unit
  Visit 2 (n=19) | 2.72 (1.50)
  Visit 3 (n=17) | 3.69 (1.97)
  Visit 5 (n=16) | 4.42 (2.55)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.05, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.18, ANOVA

8. Primary Outcome: Mean Fluorescence Intensity of Membrane Bound Tumor Necrosis Factor Alpha (mTNFα) on Neutrophil Surface
Description: Neutrophils were incubated with labeled antibody against mTNF. Flow cytometry was used to determine the mean fluorescence intensity. Greater fluorescence correlates to a greater density of membrane bound TNF.
Time Frame: Visits 2, 3, and 5 (Baseline and Weeks 4 and 12)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: fluorescence intensity unit
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
fluorescence intensity unit
  Visit 2 (n=19) | 3.49 (3.32)
  Visit 3 (n=17) | 3.55 (3.29)
  Visit 5 (n=16) | 3.75 (4.85)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.48, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.43, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.44, ANOVA

9. Primary Outcome: Mean Chemiluminescence (Area Under the Concentration-time Curve [AUC]) of Neutrophil Reactive Species Production Using Formyl-Methionyl-Leucyl-Phenylalanine (fMLP) Stimulation
Description: Using luminol as a substrate for reactive oxidants, a chemical reaction is produced resulting in photon emission (chemiluminescence). fMLP stimulation is mediated through the fMLP receptor on the cell surface. The fMLP response is only observed in primed neutrophils and response is a measure of in vivo priming. Measurements of reactive oxygen species are calculated as total chemiluminescence or the AUC.
Time Frame: Visit 2, 3, 5, and 8 (Baseline and predose at Weeks 4, 12 and 24)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: chemiluminescence units*hours
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
chemiluminescence units*hours
  Visit 2 (n=19) | 8671 (4597.18)
  Visit 3 (n=18) | 9971 (7139.36)
  Visit 5 (n=17) | 32361 (72947.87)
  Visit 8 (n=14) | 10573 (5537.06)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.313, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.083, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.092, ANOVA
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.145, ANOVA
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.398, ANOVA
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.138, ANOVA

10. Primary Outcome: Mean Chemiluminescence (AUC) of Neutrophil Reactive Species Production Using Phorbol 12-Myristate 13-Acetate (PMA) Stimulation
Description: Using luminol as a substrate for reactive oxidants, a chemical reaction is produced resulting in photon emission (chemiluminescence). PMA is a receptor-independent stimulator of the respiratory burst and the PMA response measures the total capacity of neutrophils to generate reactive oxidants. Measurements of reactive oxygen species are calculated as total chemiluminescence or the AUC.
Time Frame: Visit 2, 3, 5, and 8 (Baseline and predose at Weeks 4, 12 and 24)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: chemiluminescence units * hours
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
chemiluminescence units * hours
  Visit 2 (n=19) | 141039 (72621.95)
  Visit 3 (n=18) | 145304 (48836.93)
  Visit 5 (n=17) | 157028 (73054.72)
  Visit 8 (n=14) | 116968 (51291.31)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.467, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.250, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.060, ANOVA
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.149, ANOVA
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.061, ANOVA
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.047, ANOVA

11. Primary Outcome: Percentage of Neutrophils Positive for Propidium Iodide (PI)-Labeled Staphylococcus Aureus (S. Aureus) Uptake
Description: S. aureus were heat killed then labeled with PI and opsonized with AB serum (SAPI). S. aureus was then incubated with the neutrophils for 30 minutes at 37 degrees Celsius. The neutrophils were washed, then the percentage of cells positive for the labeled S. aureus (that is, phagocytosed) was calculated via flow cytometry. A higher percentage represented more active phagocytosis.
Time Frame: Visit 2, 3, 5, and 8 (Baseline and Weeks 4, 12 and 24)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percentage of positive neutrophils
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
percentage of positive neutrophils
  Visit 2 (n=19) | 96.59 (3.01)
  Visit 3 (n=19) | 97.47 (2.56)
  Visit 5 (n=17) | 97.53 (2.68)
  Visit 8 (n=15) | 97.25 (2.27)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.169, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.165, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.471, ANOVA
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.243, ANOVA
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.396, ANOVA
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.375, ANOVA

12. Primary Outcome: Percentage of Neutrophils Positive for Dihydrorhodamine-123 (DHR) Oxidation
Description: Phagocytosis can be measured by incubating neutrophils with PI-labeled heat killed S. aureus following incubation for 30 minutes. Neutrophils are co-incubated with DHR, which becomes oxidized by the products of the respiratory burst generated during phagocytosis. Fluorescence can then be measured by flow cytometry.
Time Frame: Visit 2, 3, 5, and 8 (Baseline and Weeks 4, 12 and 24)
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: percentage of positive neutrophils
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 19
percentage of positive neutrophils
  Visit 2 (n=19) | 99.21 (2.43)
  Visit 3 (n=19) | 99.20 (1.93)
  Visit 5 (n=17) | 99.91 (0.18)
  Visit 8 (n=15) | 99.92 (0.22)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Visit 3 versus Visit 2; Test type: Superiority or Other; p = 0.496, ANOVA
Statistical Analysis 2: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 2; Test type: Superiority or Other; p = 0.122, ANOVA
Statistical Analysis 3: Comparison: Tocilizumab 8 mg/kg; Visit 5 versus Visit 3; Test type: Superiority or Other; p = 0.070, ANOVA
Statistical Analysis 4: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 2; Test type: Superiority or Other; p = 0.135, ANOVA
Statistical Analysis 5: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 3; Test type: Superiority or Other; p = 0.082, ANOVA
Statistical Analysis 6: Comparison: Tocilizumab 8 mg/kg; Visit 8 versus Visit 5; Test type: Superiority or Other; p = 0.461, ANOVA

13. Secondary Outcome: Disease Activity Score Based on 28-Joint Count (DAS28)
Description: The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis. The index includes swollen and tender joint counts, acute phase response (erythrocyte sedimentation rate [ESR] or C-reactive protein [CRP]), and general health status. The DAS28, which uses a 28 joint count, is derived from the original DAS, which includes a 44 swollen joint count. The DAS28 scale ranges from 0 to 10, where higher scores represent higher disease activity.
Time Frame: Screening, Baseline, and Weeks 4, 8, 12, 16, 20, 24, 36, 48, and 52
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 21
score on a scale
  Screening (n=21) | 5.67 (1.22)
  Baseline (n=21) | 6.15 (1.26)
  Week 4 (n=21) | 4.90 (1.40)
  Week 8 (n=20) | 4.31 (1.64)
  Week 12 (n=20) | 3.83 (1.45)
  Week 16 (n=20) | 3.81 (1.69)
  Week 20 (n=20) | 3.92 (1.45)
  Week 24 (n=16) | 3.26 (1.49)
  Week 36 (n=12) | 3.27 (1.33)
  Week 48 (n=11) | 3.59 (1.62)
  Week 52 (n=18) | 3.58 (1.51)

14. Secondary Outcome: Percentage of Participants With Acceptable and Not Acceptable Benefit-Risk Assessments
Description: Benefit:Risk was defined at the participant level. It was considered acceptable if the DAS28 improvement represented at least a moderate European League Against Rheumatism (EULAR) response. The risks were based on the known adverse event (AE) profile of tocilizumab rather than on the actual AEs experienced by each participant
Time Frame: Weeks 12, 24, and 36
Population: ITT Population; n=number of participants analyzed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 20
percentage of participants
  Acceptable, Week 12 | 100
  Not Acceptable, Week 12 | 0
  Acceptable, Week 24 | 94
  Not Acceptable, Week 24 | 6
  Acceptable, Week 36 | 92
  Not Acceptable, Week 36 | 8

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of Screening until the End of Study which was the follow up visit after 48 Weeks of extension treatment period.
Arm/Group | Tocilizumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=21)
Neutropenia (Blood and lymphatic system disorders) | 1 — After the third Tocilizumab administration was given patient had a neutrophil count of 0.39 x 109/L. No infection was reported. when the neutrophil count reached back to 2.16 x 109/L, the event was considered to have resolved without intervention.
Pneumonia Viral (Infections and infestations) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab 8 mg/kg (N=21)
Neutropenia (Blood and lymphatic system disorders) | 2
Ear infection (Infections and infestations) | 3
Lower respiratory tract infection (Infections and infestations) | 9
Nasopharyngitis (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 4
Malaise (General disorders) | 3
Neutrophil count decreased (Investigations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Joint lock (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2
Peripheral coldness (Vascular disorders) | 2
Palpitations (Cardiac disorders) | 1
Cushingoid (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Candidiasis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Blood cholesterol increased (Investigations) | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Dysmenorrhea (Reproductive system and breast disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Heat rash (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the sponsor's intellectual property rights.